CLINICAL TRIAL: NCT05094271
Title: Is Obstructive Sleep Apnea Important in the Development of Alzheimer's Disease?
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Atul Malhotra, Professor, Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 200228
Record Dates: First submitted 2021-10-22; First posted 2021-10-26 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: OSA; Sleep Apnea; Obstructive Sleep Apnea; Alzheimer Disease
Keywords: sleep; OSA; Sleep Apnea; Obstructive Sleep Apnea; Alzheimer Disease; Sleep Disorder; Alzheimer
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Alzheimer Disease; Sleep Wake Disorders | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Masking Description: If subjects have been randomized to receive room air, subjects will have a nasal cannula with pressurized room air to avoid unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Supplemental Oxygen during PSG (Active Comparator): Subjects will be instrumented with a nasal cannula to receive 2L/min supplemental oxygen. The oxygen will be kept at a fixed rate, however, the participant will be titrated to receive a max of 4 liters per min to maintain sats >90% based on oximetry readings.
  Interventions: Other: Supplemental Oxygen
- Room Air during PSG (Placebo Comparator): Subjects will be instrumented with a nasal cannula to receive 2L/min of pressurized room air. The room air will be kept at a fixed rate, however, the participant will be titrated to receive a max of 4 liters per min to maintain sats >90% based on oximetry readings.
  Interventions: Other: Room Air
- Supplemental Oxygen for 3 Months (Experimental): Over a 12-week period, participants randomized to receive supplemental Oxygen for treatment of OSA will be contacted weekly to be asked about their adherence. Participants' adherence will also be monitored remotely through cloud-based monitoring.
  Interventions: Other: Supplemental Oxygen
- PAP Therapy for 3 Months (Experimental): Over a 12-week period, participants randomized to receive supplemental PAP therapy for treatment of OSA will be contacted weekly to be asked about their adherence. Participants' adherence will also be monitored remotely through cloud-based monitoring.
  Interventions: Device: Continuous Positive Airway Pressure Machine

INTERVENTIONS:
Other: Supplemental Oxygen — Subjects will be instrumented with a nasal cannula to receive 2L/min supplemental oxygen. The oxygen will be kept at a fixed rate, however, the participant will be titrated to receive a max of 4 liters per min to maintain sats >90% based on oximetry readings.
  Other Names: Oxygen; O2
  Arms: Supplemental Oxygen during PSG; Supplemental Oxygen for 3 Months
Device: Continuous Positive Airway Pressure Machine — Continuous positive airway pressure is a form of positive airway pressure ventilation in which a constant level of pressure greater than atmospheric pressure is continuously applied to the upper respiratory tract of a person.
  Other Names: CPAP; PAP
  Arms: PAP Therapy for 3 Months
Other: Room Air — Subjects will be instrumented with a nasal cannula to receive 2L/min pressurized room air. The room air will be kept at a fixed rate, however, the participant will be titrated to receive a max of 4 liters per min to maintain sats >90% based on oximetry readings.
  Other Names: Placebo
  Arms: Room Air during PSG

SUMMARY:
Obstructive sleep apnea (OSA) is common in older adults and has recently been implicated in pathogenesis of Alzheimer's disease (AD). Research has shown that sleep disruptions have caused memory impairment. Sleep apnea is a form of sleep disruption. We would like to examine how obstructive sleep apnea may contribute to the progression of Alzheimer's disease.

DETAILED DESCRIPTION:
Aim 1: We will assess the endotypes (mechanisms) underlying OSA in elderly individuals known to be high risk for AD (vs. non-OSA matched controls) using novel recently validated simplified techniques which do not require burdensome complex overnight experiments to assess endotypes (primary outcome loop gain). We will further assess the predicted response to O2 therapy in terms of respiratory outcomes among elderly OSA patients with varying levels of loop gain and pharyngeal collapsibility.

Hypothesis 1: A substantial proportion of high AD risk patients with OSA should be O2 responsive as predicted using pathophysiological assessments.

Aim 2: We will perform an overnight mechanistic study of oxygen therapy vs. room air in high AD risk patients with OSA (recruited from Aim 1 and others if necessary). Given the frequent intolerance of PAP in elderly patients, we anticipate that oxygen therapy may be a viable therapeutic approach in this fragile population. We will focus on respiratory outcomes (primary outcome: apnea hypopnea index) but also assess sleep dependent memory consolidation on word pairs task given the major impact in the elderly.

Hypothesis 2: O2, compared to room air, will improve OSA and neurocognitive outcomes in select elderly OSA patients at risk of AD.

Aim 3: Preclinical AD with OSA and non-OSA controls, from Aim 1 will have structural and molecular brain imaging focusing on hippocampal atrophy as a predictor of memory consolidation. We will also assess amyloid and tau in the medial temporal region as function of OSA severity and as a predictor of neurocognitive function. This aim will lay the groundwork for designing a robust clinical trial using neuroimaging outcomes.

Hypothesis 3: Impairment in memory consolidation is a function of hippocampal size in OSA patients at risk of AD.

Aim 4: We will perform a pilot randomized trial of oxygen vs. PAP therapy in OSA patients with preclinical AD.

Hypothesis 4: In preclinical AD with OSA, oxygen will be a viable therapeutic strategy to improve memory.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-85 years
2. Gender: Men or Women
3. MOCA > 26
4. Independently living and able to drive
5. OSA (AHI ≥ 15/h) or no OSA
6. Subjects must consent to waiving their right to obtain their PHS score (since the score is not yet actionable and could lead to social stress and ethical dilemmas)

Exclusion Criteria:

1. Currently smoking
2. History of COPD or asthma
3. Heart Failure Class III or IV, unstable cardiovascular disease, or uncontrolled hypertension
4. Neuromuscular Disease
5. Drowsy Driving (ESS > 18/24)
6. Inability to complete study procedures, such as questionnaire that are only available/validated in English
7. Lack of decisional capacity to provide informed consent
8. Participants in whom magnetic resonance imaging Magnetic Resonance Imaging [MRI] is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant
9. Presence of a brain tumor or lobar stroke
10. Current drug or alcohol abuse/dependence
11. Prisoners

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Loop Gain (LG) | 8 hours
  A method used to measure respiratory stability of the negative feedback chemoreflex control system using a specialized Positive Airway Pressure machine called a pCrit. The overall loop gain of the ventilatory system reflects the ratio of the ventilatory response to the disturbance that elicited the response (LG = ventilatory response/ventilatory disturbance). The higher the loop gain, the potentially more unstable the respiratory control system becomes.
Apnea Hypopnea Index | 8 hours
  The number of times a person stops breathing and periods of shallow breathing with a marked decrease in blood oxygen concentration every hour on average. A score lower than five indicates normal sleep (no sleep apnea), 5-15 indicates mild sleep apnea, 15-30 indicates moderate sleep apnea, and a score greater than 30 indicates severe sleep apnea.
Neuroimaging | 2 hours
  MRI and PET Scans. This study will examine pre-clinical AD with OSA patients using brain imaging (structural MRI and amyloid/tau PET). MRI will be conducted to provide a structural image suitable for coregistering the PET image and observing white matter integrity. The scan should take 35 minutes. These will be MPRAGE images collected using the standard ADNI protocol at the in-house 3T MRI scanner at the UCSD Altman Clinical and Translational Research Institute (ACTRI). The PET scan should take 70-90 minutes.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | 12 weeks
  A self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life.
Pittsburg Sleep Quality Index (PSQI) | 12 weeks
  A 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Insomnia Severity Index (ISI) | 12 weeks
  A 7-item self-report form to assess insomnia severity. Total score categories: 0-7 = No clinically significant insomnia, 8-14 = Subthreshold insomnia, 15-21 = Clinical insomnia (moderate severity), 22-28 = Clinical insomnia (severe).

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Sleep Research, La Jolla, California, United States

REFERENCES:
- [Derived] Holloway BM, Harding CD, DeYoung P, Kwan CG, Avetisyan L, Lui KK, Ancoli-Israel S, Banks SJ, Djonlagic I, Malhotra A. Comorbid insomnia and sleep apnea is associated with worse verbal episodic memory in older females. J Clin Sleep Med. 2025 Dec 1;21(12):2129-2138. doi: 10.5664/jcsm.11902. PMID 41025403
- [Derived] Harding CD, Holloway BM, DeYoung PN, Kwan C, Djonlagic I, Ancoli-Israel S, Banks SJ, Malhotra A. Subjective daytime sleepiness, not sleep quality or hypoxia, predicts sleep-dependent memory consolidation in a cohort of older adults. J Clin Sleep Med. 2025 Jul 1;21(7):1217-1226. doi: 10.5664/jcsm.11648. PMID 40135690